CLINICAL TRIAL: NCT01417247
Title: Renal Sympathetic Modification in Patients With Metabolic Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Director and Professor, Dept. of Cardiology, the second affiliated hospital of Chongqing Medical University, Chongqing Cardiac arrhythmias service center, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWAN-MS
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Metabolic Syndrome
Keywords: renal artery; sympathetic nerves; modification; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- renal sympathetic modification (Experimental): Renal artery ablation to modify sympathetic activity in patients with metabolic syndrome.
  Interventions: Procedure: renal sympathetic modification
- Absolute medicine therapy (No Intervention): Maintenance of anti-metabolic syndrome medications only

INTERVENTIONS:
Procedure: renal sympathetic modification — Device: THERMOCOOL® Catheter Renal sympathetic modification with a catheter-based procedure
  Other Names: renal denervation
  Arms: renal sympathetic modification

SUMMARY:
The purpose of this study is to observe the incident of composite cardiovascular events after renal sympathetic modification using THERMOCOOL® catheter in patients with metabolic syndrome, and evaluate safety and efficacy of the intervention.

DETAILED DESCRIPTION:
Metabolic syndrome is combination risk factors of serial cardiovascular and metabolic disease, included central obesity, insulin resistance, dyslipidemia, and hypertension. Basic studies suggested that sympathetic nerves over activity played an important role in the development and perpetuation of metabolic syndrome. Clinical therapies occurred by complication treatment and therapeutic life-style changes. Present study of renal ablation for sympathetic modification shows a new method to decrease sympathetic nerves activity. We assume that modifying renal sympathetic activity by ablation is effective and safe in treatment of metabolic syndrome. This trial is going to recruit 200 patients (Ablation group VS Control group = 1:1) with a follow-up duration of 3 years. Patients in ablation group will receive additional necessary medications besides expectant intervention, and patients in control group will receive appropriate medications only. We aim to observe the incident of composite cardiovascular events after renal sympathetic modification using THERMOCOOL® catheter in patients with hypertension, and evaluate safety and efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, and ≤ 75 years old of age
* abnormal metabolism: 1) body mass index (BMI) of ≥ 25 kg/m2; 2) total triglyceride (TG) of ≥ 1.70mmol/l (150mg/dl); 3) high density lipoprotein- cholesterol (HDL-C) of male <0.91mmol/l (35mg/dl), and of female <1.01mmol/l (39mg/dl); 4)fasting blood glucose 6.1mmol/l (110mg/dl), or glucose tolerance test of 2 hours ≥ 7.8 mmol/l (140mg/dl); 5), or history of diabetes mellitus
* estimated glomerular filtration rate (eGFR) of ≥ 45mL/min
* is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

* secondary hypertension
* type 1 diabetes mellitus
* estimated glomerular filtration rate (eGFR) of < 45mL/min
* has the history of renal restenosis or renal stents implantation
* has experienced AMI (old myocardial infarction is not excluded), unstable angina pectoris, cerebrovascular accidents, and alimentary tract hemorrhage within 3 months
* patients with sick sinus syndrome
* pregnant women
* mental disorders
* patients that have allergy to contrast agent
* patients that do not go with follow-up
* others such as researcher considers it is not appropriate to be included into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
composite cardiovascular events (myocardial infarction, heart failure, sudden death, cardiogenic death) | three years

SECONDARY OUTCOMES:
effect of glucose and lipid metabolism, and blood pressure variability | three years

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China